CLINICAL TRIAL: NCT04860388
Title: Comparison of the Gingival Thickness, Keratinized and Attached Gingival Widths of Unilateral Labially and Palatally Impacted Maxillary Canines Erupted by Closed Eruption Technique
Brief Title: Gingival Thickness of Impacted Maxillary Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nazli Zeynep Alpaslan Yayli, PhD, DDA, Assistant professor, Yuzuncu Yil University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 29.05.2019/10
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Impacted Canines; Orthodontic Treatment; Gingival Thickness
Keywords: Impacted Canine; Closed Eruption Technique; Gingival Thickness; Keratinized Gingival Width; Attached Gingival Width

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral labially impacted maxillary canines (Active Comparator): Distalization of the maxillary molars and/or protrusion of the maxillary and mandibular incisors made for creating sufficient space for impacted maxillary canines. After sufficient space for impacted maxillary permanent canine was obtained combine surgical-orthodontic treatment was performed via closed eruption technique. When the crown of the maxillary impacted canine was fully visible in the mouth, its bracket was inserted, and aligned within the dental arch. Posttreatment plaque index, gingival index, gingival bleeding index, probing depth, keratinized and attached gingival width and gingival thickness measurements of the impacted canines and controls were performed. The periodontal health of labially impacted maxillary canines compared with the contralateral canines that served as control teeth.
  Interventions: Procedure: closed eruption technique
- unilateral palatally impacted maxillary canines (Active Comparator): Distalization of the maxillary molars and/or protrusion of the maxillary and mandibular incisors made for creating sufficient space for impacted maxillary canines. After sufficient space for impacted maxillary permanent canine was obtained combine surgical-orthodontic treatment was performed via closed eruption technique. When the crown of the maxillary impacted canine was fully visible in the mouth, its bracket was inserted, and aligned within the dental arch. Posttreatment plaque index, gingival index, gingival bleeding index, probing depth, keratinized and attached gingival width and gingival thickness measurements of the impacted canines and controls were performed. The periodontal health of palatally impacted maxillary canines compared with the contralateral canines that served as control teeth.
  Interventions: Procedure: closed eruption technique

INTERVENTIONS:
Procedure: closed eruption technique — The impacted teeth treated with closed eruption technique firstly. Orthodontic traction started a week later the sutures were removed. When the crown of the maxillary impacted canine was fully visible in the mouth, its bracket was inserted, and aligned within the dental arch using double-arch technique. Posttreatment plaque index, gingival index, gingival bleeding index, probing depth, and keratinized and attached gingival width and gingival thickness measurements of the impacted canines and controls were performed. The measurements compared with the contralateral canines that served as control teeth.

SUMMARY:
This study was conducted to compare the periodontal health of labially and palatally impacted maxillary canines with similar mesio-distal displacement, perpendicular distance, and angulation, and to compare them with the contralateral canines that served as control teeth. Two null hypothesis were tested: (1) there are no differences in attached and keratinized gingival widths and gingival thickness between impacted teeth and controls, and (2) there are no differences in attached and keratinized gingival widths and gingival thickness of labially and palatally impacted canines.

DETAILED DESCRIPTION:
When a tooth is embedded in the alveolar bone and fails to erupted into the oral cavity within the expected time, dental impaction occurs. Maxillary canine impaction has been observed more frequently in the palatal position than labial position, and unilaterally than bilaterally. Treatment of these teeth, which consitute a transition between the anterior and posterior dental segments and therefore have a great of importance both from functional and aesthetic point of view, is recommended rather than extraction.

Many complications that have been reported to be faced during the surgical exposure and orthodontic alignment of the impacted teeth are devitalization, external root resorption, damage to adjacent teeth, marginal bone loss, re-exposure of the tooth, and gingival recession. Gingival recession is the apical migration of the gingival margin beyond the cementoenamel junction, resulting in the clinical exposure of the root surface. The term gingival biotype is generally used to describe the thickness of the gingiva in faciolingual/faciopalatinal direction.

Although a large number of existing studies in the broader literature have examined the periodontal health of labially and palatally impacted maxillary canines seperately, limited number of studies compared the labially and palatally maxillary impacted canines. Since one of the factors affecting the posttreatment periodontal health is the initial vertical and horizontal position of the impacted teeth, these studies were observed not provided any information about the pretreatment mesio-distal displacement, perpendicular distance and angulation of the impacted maxillary canines. At this point, this study was conducted to compare the periodontal health of labially and palatally impacted maxillary canines with similar mesio-distal displacement, perpendicular distance, and angulation, and to compare them with the contralateral canines that served as control teeth. Two null hypothesis were tested: (1) there are no differences in attached and keratinized gingival widths and gingival thickness between impacted teeth and controls, and (2) there are no differences in attached and keratinized gingival widths and gingival thickness of labially and palatally impacted canines.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were no previous functional orthopaedic and/or fixed orthodontic treatment, complete permanent dentition, aged between 13 and 20 years old at the begining of the treatment, no systemic problems and related medications, good oral hygiene, no gingival inflammation and periodontal diseases, unilateral labially or palatally impacted maxillary canines, indication of surgical uncovering of the impacted maxillary canine using closed eruption technique, presence of normally positioned contralateral maxillary canine, and complete good quality pretreatment and posttreatment records.

Exclusion Criteria:

* Subjects who had fixed orthodontic treatment with teeth extraction, missing teeth adjacent to the canine, and significant distortion between the left and right half jaws in the initial panoramic radiographs were excluded from the study.

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Gingival Thickness measurement (mm) | 6 months after the completion of orthodontic treatment
  The gingival thicknesses of the impacted canines and controls measured along the long axis of the midbuccal surfaces of teeth under topical anaesthesia at two points: apical to the free gingival margin and coronal to the mucogingival junction. A 15-mm endodontic spreader was perpendicularly positioned to the long axis of the measurement points and gently inserted into the soft tissue until feeling the resistance of alveolar bone. Then, the endodontic spreader was carefully removed and the penetration depth between the tip of the endodontic spreader and silicon stopper was registered using a digital caliper with 0.01-mm sensivity

SECONDARY OUTCOMES:
keratinized gingival width measurement (mm) | 6 months after the completion of orthodontic treatment
  The keratinized (distance from the gingival margin to the mucogingival junction) gingival width measurements of the impacted canines and controls performed, clinically, parallel to the long axis of teeth at the midbuccal root surfaces .
attached gingival width measurement (mm) | 6 months after the completion of orthodontic treatment
  The attached (distance from the gingival groove base to the mucogingival junction) gingival width measurements of the impacted canines and controls performed, clinically, parallel to the long axis of teeth at the midbuccal root surfaces.
plaque index score (0-3) | 6 months after the completion of orthodontic treatment
  Plaque index of the impacted canines and controls were measured from the 6 surfaces of each tooth. The plaque index score of each tooth was calculated with Silness-Loe plaque index by dividing the total value by 6.
  0: absence of microbial plaque
  1. Thin film of microbial plaque along the free gingival margin
  2. moderate accumulation with plaque in the sulcus
  3. large amount of plaque in sulcus or pocket along the free gingival margin
gingival index score (0-3) | 6 months after the completion of orthodontic treatment
  The gingival index of the impacted canines and controls were measured from the 6 surfaces of each tooth. The gingival index score of each tooth was calculated with Silness-Loe gingival indeks by dividing the total value by 6.
  0: Normal gingiva
  1. Mild inflammation: slight change in color, slight oedema, no bleeding on probing
  2. Moderate inflammation: redness, oedema and glazing, bleeding on probing
  3. Severe inflammation: marked redness and oedema, ulceration, tendency to spontaneous bleeding
gingival bleeding index score (percentage) | 6 months after the completion of orthodontic treatment
  Bleeding on probing scores of the impacted canines and controls were measured by Ainamo and Bay's gingival bleeding index from 6 surfaces of each tooth. If there is bleeding after probing, it is recorded as +, if there is no bleeding it is recorded as _. Gingival bleeding index is calculated as a percentage of affected sites.
probing depth measurement (mm) | 6 months after the completion of orthodontic treatment
  Probing depth (PD) (distance from gingival margin to gingival pocket base) of the impacted canines and controls were measured with a probe in 6 regions of each tooth and recorded as mm. measured with a probe in 6 regions of each tooth and recorded as mm.

CONTACTS AND LOCATIONS:
Overall Officials: Nazli Zeynep Alpaslan Yayli, PhD, Principal Investigator — Yuzuncu Yil University; Yesim Kaya, PhD, Study Chair — Ankara Yildirim Beyazıt University; Saadet Cinarsoy Cigerim, PhD, Study Chair — Yuzuncu Yil University
Locations (1):
- Nazli Zeynep Alpaslan Yayli, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mummolo S, Nota A, De Felice ME, Marcattili D, Tecco S, Marzo G. Periodontal status of buccally and palatally impacted maxillary canines after surgical-orthodontic treatment with open technique. J Oral Sci. 2018 Dec 27;60(4):552-556. doi: 10.2334/josnusd.17-0394. Epub 2018 Jul 9. PMID 29984786